CLINICAL TRIAL: NCT05571332
Title: Efficacy and Safety of Avatrombopag Combined With IST for the Treatment of HAAA and SAA With Abnormal Liver Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021008-EC-1(2)
Record Dates: First submitted 2022-08-28; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-08

CONDITIONS: Aplastic Anemia
Keywords: Avatrombopag; aplastic anemia; abnormal liver function; hepatitis
MeSH Terms: conditions — Anemia, Aplastic; Liver Diseases; Hepatitis | interventions — avatrombopag; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatrombopag+CsA+ p-ATG (Experimental): Patients received p-ATG for 5 consecutive days (day 1-5), at a dose of 20 mg/kg/day. CSA is started at 3 mg/kg orally in two doses. Concentrations maintained at 200-250 ng/ml to achieve maximum efficacy and then tapered by 25 mg every 3 months; Avatrombopag: 40 mg orally once daily for a total of 12 weeks. A total of 39 patients were expected to be included.
  Interventions: Drug: Avatrombopag 20 MG Oral Tablet

INTERVENTIONS:
Drug: Avatrombopag 20 MG Oral Tablet — p-ATG and CsA in combination with Avatrombopag to treat
  Other Names: porcine ATG; Cyclosporine(CsA)

SUMMARY:
This is a multicenter, single-arm clinical study. The objective was to evaluate the efficacy and safety of Avatrombopag combined with IST in very/sever aplastic anemia patients with abnormal liver function or HAAA patients treated for the first time. The design was: Patients received p-ATG for 5 consecutive days (day 1-5), at a dose of 20 mg/kg/day. Cyclosporine 3 mg/kg orally in two divided doses, with cyclosporine trough concentrations maintained at 200-250 ng/ml for 3 months to achieve maximum efficacy, and Avatrombopag, which was administered in the dose of 40 mg orally once daily for a total of 12 weeks. Thirty-nine patients are expected to be enrolled in this study. Evaluation endpoint: complete response rate at 12 weeks of treatment.

DETAILED DESCRIPTION:
This is a multicenter, single-arm clinical study to evaluate the efficacy and safety of Avatrombopag combined with IST as the first-line regimen for aplastic anemia. The patients are diagnosed as hepatitis associated with very sever/sever aplastic anemia(V/SAA) or V/SAA with abnormal liver function before treatment.

Patients received p-ATG for 5 consecutive days (day 1-5), at a dose of 20 mg/kg/day. CSA is started at 3 mg/kg orally in two doses. Concentrations maintained at 200-250 ng/ml to achieve maximum efficacy and then tapered by 25 mg every 3 months; Avatrombopag: 40 mg orally once daily for a total of 12 weeks. A total of 39 patients were expected to be included.Complete response rate at 12 weeks of treatment and adverse events are the evaluation endpoint.Secondary study endpoints were: ORR at 12 , CRR and ORR at 24 weeks, survival, and clonal evolution in follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. patients with V/SAA with a definite diagnosis.
2. age between 18-70 years, male or female.
3. Subjects must complete all screening assessments as outlined in the trial protocol.
4. Able to swallow or administer the drug orally.
5. No prior application of TPO receptor agonists (including Thrombopoietin, Eltrombopag, Hetrombopag, etc.) or application of TPO receptor agonists for treatment with ≤ 5 total doses and ≤ 7 days of TPO receptor agonist drugs such as Eltrombopag, Hetrombopag, etc.
6. Diagnosis as HAAA or abnormal liver function. ALT and AST more than 1.5 times of upper limit.
7. Informed consent must be signed prior to the start of all specific study procedures, in consideration of the patient's condition, or by a member of the patient's immediate family if the patient's signature is not conducive to the treatment of the condition.

Exclusion Criteria:

1. Known diagnosis of congenital hematopoietic failure disorders (e.g. Fanconi anemia) and other causes of allogeneic cytopenias and bone marrow hypoproliferative disorders (e.g. hemolytic PNH, hypoproliferative MDS/AML, autoantibody-mediated allogeneic cytopenias, etc.);
2. Patients with uncontrolled bleeding and/or infection despite standard treatment.
3. Patients with previous history of hematopoietic stem cell transplantation; previous history of thrombosis.
4. Patients with concurrent malignancy or potential cancer on immunosuppressive therapy.
5. Those who are considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
CR rate at 12 weeks of treatment | 12 weeks of treatment
  Percentage of the total number of patients receiving treatment who received a complete response at 12 weeks of treatment
ncidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading at 12 weeks of treatment | 12 weeks of treatment
  Incidence of Treatment-Emergent AE by CTCAE

SECONDARY OUTCOMES:
OR rate at 12 weeks of treatment | 12 weeks of treatment
  Percentage of the total number of patients receiving treatment who received a response at 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wenrui Yang, Study Director — Anemia Therapeutic center
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
You can ask for the researcher after completing the experiment
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Follow-up and publication of the paper are planned for December 2024
Access Criteria: After the paper is written and published

REFERENCES:
- [Result] Young NS, Kaufman DW. The epidemiology of acquired aplastic anemia. Haematologica. 2008 Apr;93(4):489-92. doi: 10.3324/haematol.12855. No abstract available. PMID 18379007
- [Result] Scheinberg P. Activity of eltrombopag in severe aplastic anemia. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):450-456. doi: 10.1182/asheducation-2018.1.450. PMID 30504345